CLINICAL TRIAL: NCT04661800
Title: Prevalence and Characteristics of Alterations in Olfactory and Taste Function in Patients With Cardiac Amyloidosis and Nutritional Impact: Multicenter Cross-sectional Study
Brief Title: Study of Olfactory Disorders in Patients With Cardiac Amyloidosis
Acronym: AMYLODOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP200835
Record Dates: First submitted 2020-11-19; First posted 2020-12-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Amyloidosis; Cardiac Amyloidosis; Olfactory Loss; Hyposmia; Dysosmia; Smell Disorders; Taste Disorders
Keywords: Amyloidosis; cardiac amyloidosis; olfactory loss; hyposmia; dysosmia; smell disorders; taste disorders
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial; Anosmia; Olfaction Disorders; Taste Disorders

STUDY DESIGN:
Intervention Model Description: Model description: Successive monocentric cross-sectional study on the screening of smell and taste disorders carried out as part of a cardiology hospitalization programmed for the cardiology follow-up of his pathology in a population of patients diagnosed with AC. All subjects will have an ENT check-up including: an ENT examination with a nasal endoscopy, an evaluation of the olfactory function by Sniffin's stick tests (test which consists of smelling smelling pens) an evaluation of taste (test which consists of discriminating between acid, bitter, sweet and salty using blotting papers placed on the tongue). Nutritional status will be assessed by a mini-questionnaire, measurement of weight, brachial circumference and tricipital skin fold, calculation of body mass index (BMI), orosomucoid dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test de bâton de Sniff (Other): Cohorte
  Interventions: Other: Sniffin's stick test

INTERVENTIONS:
Other: Sniffin's stick test — The sniffin's stick test is a three-part test consisting of smelling odor pens: 1) determining a detection threshold, 2) discriminating ability, 3) ability to identify odors. It lasts about 30 minutes, is achievable in the room.

SUMMARY:
Amyloidosis is a disease caused by the continuous accumulation of fibrillary proteins in the extracellular matrix causing the architecture of different organs to be disrupted. The prevalence of the disease increases with age. The two most common forms are light chain amyloidosis (AL) and transthyretin (TTR). TTR amyloidosis may be hereditary (m-TTR, or mutated) or age-related (WT-TTR, or wild). The latter is also called senile amyloidosis. In all these forms, cardiac impairment is common and leads the patient to consult/or be referred to a cardiological center unfortunately often too late when the prognosis is directly related to the severity of the heart attack. The description/discovery of clinical signs prior to heart disease is important to improve the detection and diagnosis of early forms of cardiac amyloidosis (CA). For example, an infiltration of the carpal tunnel synovial by amyloid deposits is observed in some patients, 5 years before the onset of signs of heart failure and is the only warning sign of the disease known to date. We also showed in a previous study that patients had more severe and earlier impairment of hearing function than expected by age and gender.

Objective The main objective is to define the prevalence and severity of smell and taste disorders in a population of patients with cardiac amyloidosis (3 types of mutated or wild AL amyloidosis and TTR).

The main endpoint is to determine the number of patients with impaired smell and taste's functions in a population of patients diagnosed with cardiac amyloidosis (3 types of mutated (hereditary) or senile wild amyloidosis (3 types of AL amyloidosis and TTR).

Method Successive monocentric cross-sectional study on the screening of smell and taste disorders carried out as part of a cardiology hospitalization programmed for the cardiology follow-up of his pathology in a population of patients diagnosed with AC.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Affiliated with Social Security
* Patient who was informed of the study and signed a free and informed consent
* Patients diagnosed with AC

Exclusion Criteria:

* - Refusal to participate in the study
* Patient who does not speak or understand French
* History of chronic rhino sinusitis with or without polyps
* A history of counter-indicating the completion of nasal endoscopy (repeated epistaxis, obstructive naso-sinusal tumors, choanal imperforation)
* History of major craniofacial trauma resulting in loss of smell
* Known history of Parkinson's disease or Alzheimer's disease
* Antecedent of ENT radiotherapy
* History of chemotherapy
* Patient under guardianship, curatorship or legal protection
* Patient on AME
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of smell and taste disorders in a population of patients with cardiac amyloidosis | at inclusion day
Severity of smell and taste disorders in a population of patients with cardiac amyloidosis, evaluated with Sniffin's stick tests score (score/48) | at inclusion day

SECONDARY OUTCOMES:
Date of onset of smell and taste disorder (month/years) compared with date of onset of cardiological symptoms and cardiac amyloidosis, based on declarative assessment | at inclusion day
TDI scores of Sniffin's stick test compared to Sniffin's stick test TDI scores of age and gender-matched subjects | at inclusion day
correlation between type of amyloidosis (AL, TTR mutated and wild type) and Sniffin's stick test TDI's score (/48) | at inclusion day
Correlation between severity of cardiac amyloidosis and and Sniffin's stick test TDI's score (/48). Severity of cardiac amyloidosis is evaluated by clinical characteristics (NYHA, Heart rate (bpm), Systolic Blood Pressure (mmHg), Diastolic Blood Pressure | at inclusion day
Correlation between nutritional depletion and Sniffin's stick test TDI scores (/48). Nutritional depletion is evaluated by BMI (Body mass index kg/m2), brachial circumference (cm), tricipital fold (mm), orosomucoid g/L | at inclusion day

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION